CLINICAL TRIAL: NCT07339579
Title: Evaluation of the Effects of Root Canal Sealers on Postoperative Pain and Radiographic Healing in Patients With Apical Periodontitis
Brief Title: Sealers in Chronic Apical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Aliye Kamalak, Associate Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSU-SEALER-AP-2024; 51 (22/07/2024) (Other Grant/Funding Number: HRU Ethics Committee Approval)
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Apical Periodontitis; Postoperative Pain; Periapical Healing
Keywords: Root Canal Sealer; AH Plus; MTA Fillapex; Sealapex; Root Canal Treatment; Periapical Index; Cone-Beam Computed Tomography; Postoperative Pain; Endodontics
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative | interventions — Sealapex; TheraCal

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of three parallel intervention groups according to the root canal sealer used during treatment.
Who Masked: Outcomes Assessor
Masking Description: Radiographic and CBCT images were anonymized and evaluated by independent examiners who were blinded to the intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sealapex Group (Experimental): Participants received standardized single-visit root canal treatment using Sealapex as the root canal sealer during obturation.
  Interventions: Procedure: Root Canal Treatment With Sealapex
- MTA Fillapex Group (Experimental): Participants received standardized single-visit root canal treatment using MTA Fillapex as the root canal sealer during obturation.
  Interventions: Procedure: Root Canal Treatment With MTA Fillapex
- AH Plus Group (Experimental): Participants received standardized single-visit root canal treatment using AH Plus as the root canal sealer during obturation.
  Interventions: Procedure: Root Canal Treatment With AH Plus

INTERVENTIONS:
Procedure: Root Canal Treatment With Sealapex — Root canal treatment was performed under standardized clinical conditions, and canals were obturated using gutta-percha with Sealapex (calcium hydroxide-based sealer).
  Arms: Sealapex Group
Procedure: Root Canal Treatment With MTA Fillapex — Root canal treatment was performed under standardized clinical conditions, and canals were obturated using gutta-percha with MTA Fillapex (MTA-containing salicylate resin-based sealer).
  Arms: MTA Fillapex Group
Procedure: Root Canal Treatment With AH Plus — Root canal treatment was performed under standardized clinical conditions, and canals were obturated using gutta-percha with AH Plus (epoxy resin-based sealer).
  Arms: AH Plus Group

SUMMARY:
This clinical study evaluated whether different root canal sealers influence postoperative pain and early periapical healing in patients with apical periodontitis. A total of 72 adult patients with single-rooted teeth diagnosed with chronic apical periodontitis received standardized root canal treatment and were randomly assigned to one of three commonly used sealers: AH Plus, MTA Fillapex, or Sealapex.

Postoperative pain was recorded using a verbal pain rating scale immediately after treatment and at 24 and 72 hours. Periapical healing was assessed at baseline and after six months using periapical radiographs and cone-beam computed tomography (CBCT).

The purpose of this study was to determine whether the type of root canal sealer affects patient comfort after treatment and the early healing of periapical tissues. Understanding these outcomes may help clinicians choose appropriate materials and better inform patients about expected pain and healing after root canal therapy.

DETAILED DESCRIPTION:
This study was designed as a single-center, randomized, controlled clinical trial to compare the effects of three different root canal sealers on postoperative pain and radiographic periapical healing in patients with apical periodontitis.

A total of 72 patients aged 18-65 years with single-rooted anterior or premolar teeth diagnosed with chronic apical periodontitis were enrolled. Patients with systemic diseases beyond ASA I-II status, previous endodontic treatment, root fractures, severe canal curvature, open apices, or recent use of antibiotics or analgesics were excluded to ensure standardization.

After obtaining informed consent, participants were randomly allocated into three equal groups according to the sealer used for root canal obturation: Sealapex (calcium hydroxide-based sealer), MTA Fillapex (MTA-containing salicylate resin-based sealer), or AH Plus (epoxy resin-based sealer). All root canal treatments were performed in a single visit under rubber dam isolation by the same experienced endodontist to eliminate inter-operator variability.

Root canals were prepared using a standardized nickel-titanium instrumentation system and irrigated with sodium hypochlorite and EDTA according to a uniform protocol. Obturation was completed using the lateral condensation technique with gutta-percha and the assigned sealer. Permanent composite restorations were placed after obturation.

Postoperative pain was assessed using the Verbal Rating Scale (VRS) immediately after treatment and at 24 and 72 hours. Patients were instructed not to use analgesics unless severe pain occurred.

Radiographic evaluation of periapical healing was performed using periapical radiographs and cone-beam computed tomography (CBCT) at baseline and at the 6-month follow-up. Healing was assessed using the Periapical Index (PAI) and three-dimensional CBCT evaluation to detect early changes in lesion size and bone repair.

The primary objective of the study was to compare postoperative pain levels among the three sealer groups. Secondary objectives included evaluation of early periapical healing using both two-dimensional and three-dimensional imaging methods.

This study aimed to clarify whether sealer composition influences short-term clinical outcomes when root canal treatment is performed under standardized conditions. The findings may contribute to evidence-based material selection and improved patient counseling regarding postoperative pain and healing expectations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Patients diagnosed with apical periodontitis
* Presence of a single-rooted anterior or premolar tooth with a radiographically visible periapical lesion
* Systemically healthy individuals classified as ASA I or ASA II
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Teeth with root fractures, external resorption, or open apices
* Calcified canals or severely curved root canals (>30°)
* Periodontal pocket depth greater than 3 mm
* Pregnancy
* Use of antibiotics or analgesics within the previous 7 days
* History of previous endodontic treatment or retreatment in the study tooth
* Presence of systemic conditions that could affect healing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity Assessed by Verbal Rating Scale (VRS) | Immediately after treatment, 24 hours, and 72 hours after root canal treatment
  Postoperative pain intensity was evaluated using the Verbal Rating Scale (VRS). Patients were asked to verbally rate their pain according to the following categories:
  0 = no pain, 1 = mild pain, 2 = moderate pain, and 3 = severe pain.

SECONDARY OUTCOMES:
Periapical Healing Assessed by Cone-Beam Computed Tomography (CBCT) | Baseline and 6 months after treatment
  Periapical healing was evaluated using cone-beam computed tomography (CBCT). CBCT images were analyzed to assess changes in periapical lesion size and bone healing by comparing baseline and follow-up scans.
  Healing was determined based on reduction or resolution of periapical radiolucency, assessed in coronal, sagittal, and axial sections, and supported by three-dimensional reconstruction.
  Image evaluation was performed by blinded examiners using standardized criteria.
Periapical Healing Assessed by Periapical Index (PAI) | Baseline and 6 months after treatment
  Periapical healing was assessed using the Periapical Index (PAI) based on standardized periapical radiographs.
  Radiographic findings were scored according to the five-point PAI scale as follows:
  1. = normal periapical structures,
  2. = small changes in bone structure,
  3. = changes in bone structure with some mineral loss,
  4. = periodontitis with a well-defined radiolucent area, and
  5. = severe apical periodontitis with exacerbating features.
  Changes in periapical status were evaluated by comparing baseline and 6-month follow-up images. Radiographic assessments were performed by blinded examiners using standardized evaluation criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Aliye Kamalak, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sutcu İmam University, Faculty of Dentistry, Kahramanmaraş, onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No